CLINICAL TRIAL: NCT01966081
Title: Consumption of Fatty Acids, Metabolism of Adipose Tissue and Risk of Colorectal Cancer: AGARIC Case Control Study
Brief Title: AGARIC Case Control Study
Acronym: AGARIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel
Other Study IDs: Bonithon hors AOI 2008
Record Dates: First submitted 2013-10-10; First posted 2013-10-21 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: First Recently-diagnosed Colorectal Cancer
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cases (Other)
  Interventions: Other: Blood sample; Other: tissue samples from abdominal subcutaneous adipose
- controls (Other)
  Interventions: Other: Blood sample; Other: tissue samples from abdominal subcutaneous adipose

INTERVENTIONS:
Other: Blood sample
Other: tissue samples from abdominal subcutaneous adipose

SUMMARY:
The aim of the study is to establish the existence of a relationship between the dietary intake of polyunsaturated fatty acids (PUFA) and the risk of colorectal cancer in humans, using 2 reliable and complementary biomarkers: the fatty acid-composition of lipids of the abdominal subcutaneous adipose tissue and the fatty acid composition of erythrocyte phospholipids.

ELIGIBILITY:
Inclusion Criteria:

CASES

* Patients aged ≥ 45 years
* with a first recently-diagnosed colorectal cancer
* due to undergo elective surgical resection with curative intent (in practice, stage I, II, III or IV if there was only one hepatic nodule that was resected with curative intent) in one of the 5 following digestive surgery units: CHU de Dijon, CHU de Nancy, CHU de Strasbourg, CHU de Reims et CHU and Besançon.
* who have given their informed consent

CONTROLS

* Patients aged ≥ 45 years
* due to undergo surgery for a benign abdominal disease (sigmoid diverticulitis, appendectomy, hiatal hernia …)
* matched for abdominal site with cases for age (± 3 years), sex and hospital
* Who have given their informed consent

Exclusion Criteria:

CASES

* pre-operative anticancer treatment (chemo or radiotherapy)
* existence of visceral metastases except a single hepatic nodule resected with curative intent
* familial adenomatous polyposis and HNPCC syndrome (when suspected: inclusion after complementary tumor phenotype study: screening for microsatellite instability and/or immunohistochemistry study of the expression of DNA mismatch repair proteins.
* known inflammatory disease of the intestine (ulcerative colitis, Crohn's disease)
* personal history (recent or not) of colorectal cancer
* emergency treatment for the presenting complication (perforation, occlusion…)
* significant modification in dietary habits during the previous three months
* other evolving neoplastic disease
* psychic state incompatible with understanding the modalities and the aims of the study (notably patients under guardianship)
* pregnant or breast-feeding women

CONTROLS

* personal history of cancer or adenomatous colorectal polyps,
* emergency intervention
* known inflammatory disease of the intestine (ulcerative colitis, Crohn's disease)
* personal history (recent or not) of colorectal cancer
* emergency treatment for the presenting complication (perforation, occlusion…)
* significant modification in dietary habits during the previous three months
* evolving neoplastic disease
* psychic state incompatible with understanding the modalities and the aims of the study (notably patients under guardianship)
* pregnant or breast-feeding women

Min Age: 45 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 551 (Actual)
Dates: Start 2008-09-15 (Actual); Primary Completion 2011-06-15 (Actual); Study Completion 2011-06-15 (Actual)

PRIMARY OUTCOMES:
Measure of polyunsaturated fatty acids in adipose tissue lipids. | baselines

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - CHU Jean Minjoz, Besançon
  - CHU Dijon, Dijon
  - Hôpital Robert Debré, Reims
  - Hôpital Hautepierre, Strasbourg
  - Hôpital de BRABOIS, Vandœuvre-lès-Nancy

REFERENCES:
- [Result] Cottet V, Vaysse C, Scherrer ML, Ortega-Deballon P, Lakkis Z, Delhorme JB, Deguelte-Lardiere S, Combe N, Bonithon-Kopp C. Fatty acid composition of adipose tissue and colorectal cancer: a case-control study. Am J Clin Nutr. 2015 Jan;101(1):192-201. doi: 10.3945/ajcn.114.088948. Epub 2014 Nov 12. PMID 25527763